CLINICAL TRIAL: NCT07189000
Title: A Patient-centered Prehabilitation Program to Enhance Postoperative Recovery in Patients With Malignant Cancer
Brief Title: Patient-centered REhabilitation Program to Advance REcovery
Acronym: PREPARE-CAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Eunji Ko, Clinical Assistant Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREPARE-CAN
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Frailty; Prehabilitation
Keywords: prehabilitation; frailty; cancer
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RH group (Experimental): Participants receive an app-based, patient-centered prehabilitation program from randomization until surgery (no extra clinic visits). The program includes weekly home six-minute walk tests (6MWT) logged in the app, brief daily check-ins (exercise performed, simple nutrition targets, mood/stress), push reminders, and short educational video/handout content. Safety prompts and validity checks (continuous 6 minutes, pause limits, outlier flags) are embedded in the app.
  All on-site assessments are aligned with routine care: preoperative-day in-hospital testing (primary 6MWD, plus grip/TUG/HADS; InBody via fee-free pathway where available) and one routine postoperative outpatient visit (3 or 6 months; site-standard) for follow-up secondary measures. Usual perioperative care is provided per site ERAS practice.
  Interventions: Behavioral: App-based prehabilitation program
- UC group (Active Comparator): Participants receive standard perioperative care per each site's ERAS-consistent routine (preoperative counseling/education, routine mobilization). No study app is provided and no remote 6MWT logging is required. For outcomes collection only, participants undergo the same preoperative-day in-hospital assessment (primary 6MWD, plus grip/TUG/HADS; InBody via fee-free pathway where available) and one routine postoperative outpatient visit (3 or 6 months; site-standard). No additional study-specific clinic visits are required.
  Interventions: Other: Usual care (ERAS-standard perioperative care)

INTERVENTIONS:
Behavioral: App-based prehabilitation program — A lightweight mobile/web application delivering a patient-centered prehabilitation program from randomization until surgery. Features include: weekly home six-minute walk tests (6MWT) logged in the app; brief daily check-ins for exercise performed, simple nutrition targets, and mood/stress; push reminders; short educational video/handout content; and CSV export for analysis. The app provides standardized instructions and safety prompts for the home 6MWT and basic validity checks (continuous 6 minutes, pause limits, outlier flags). No additional study-specific clinic visits are required beyond routine preoperative admission and one routine postoperative outpatient visit.
  Arms: RH group
Other: Usual care (ERAS-standard perioperative care) — Standard perioperative counseling/education and routine mobilization per institutional ERAS practice. No study app is provided and no remote 6MWT logging is required. Outcome assessments are collected at routine preoperative admission (including in-hospital 6MWT per protocol) and at one routine postoperative outpatient visit (≈3 or 6 months per unified site policy). No additional study-specific clinic visits are required.
  Arms: UC group

SUMMARY:
The goal of this clinical trial is to learn whether an app-based, patient-centered prehabilitation program improves preoperative functional capacity in adults scheduled for elective cancer surgery. The main questions it aims to answer are:

Does the program increase the six-minute walk distance (6MWD) measured on the preoperative day (within 24-48 hours before surgery)?

Compared with usual care, does the program improve preoperative adherence to home 6MWT practice and patient-reported anxiety/depression (HADS)?

Researchers will compare an app-based prehabilitation program to usual care to see if the program improves preoperative functional capacity.

Participants will:

Use a study app to perform weekly home six-minute walk tests (6MWT) and complete brief daily check-ins (exercise, nutrition, psychological status) before surgery.

Attend routine preoperative admission (no extra visit) for in-hospital 6MWT (primary endpoint) and brief assessments (grip strength, Timed Up & Go, HADS, skeletal muscle mass by InBody where available/fee-free).

Attend one routine postoperative outpatient visit at 3 or 6 months (site-standard timing) for follow-up assessments.

No additional study-specific clinic visits are required outside usual care.

DETAILED DESCRIPTION:
Overview and Rationale This multicenter, pragmatic, parallel-group randomized trial evaluates a minimal-cost, app-based, patient-centered prehabilitation program for adults undergoing elective cancer surgery. The intervention focuses on home feasibility and adherence without additional clinic visits. The single prespecified primary endpoint is defined in the Outcome Measures module. Secondary measures are collected with low or no cost (research staff-administered functional tests, app surveys/logs, and fee-free body composition where available). The design reflects three principles: (i) patient self-management supported by simple digital tools, (ii) multimodal content (exercise, nutrition, psychological support), and (iii) streamlined follow-up aligned with routine care.

Study Design and Setting Randomized (1:1), parallel assignment, open-label; outcome assessors for in-hospital functional testing will be masked when feasible. Three university hospitals participate under a common SOP and centralized coordination. Total planned enrollment is 60 participants.

Interventions

App-based prehabilitation (Experimental): Participants receive access to a lightweight mobile/web app that provides weekly prompts to perform a home six-minute walk test (6MWT), brief daily check-ins (exercise performed, simple nutrition targets, mood/stress), push reminders, and basic guidance content. The app logs attempts, completion, and distance input (or pedometer/GPS-assisted estimate when available) and allows secure CSV export for analysis.

Usual care (Control): Standard perioperative education and care per site ERAS practice; no study app.

No additional study-specific clinic visits are required. All on-site assessments are scheduled to coincide with routine preoperative admission and one routine postoperative outpatient visit (either ~3 or ~6 months, unified across sites).

Assessment Schedule (condensed, aligned to routine care)

Remote preoperative phase: Weekly home 6MWT and daily check-ins via the app until surgery (participants receive standardized instructions and safety prompts within the app).

Preoperative day (in hospital): Standardized in-hospital 6MWT on a measured indoor course; research staff administer grip strength using a calibrated hand dynamometer and the Timed Up & Go (TUG); Hospital Anxiety and Depression Scale (HADS) via app or paper; skeletal muscle mass by bioimpedance (InBody) only through fee-free pathways available at the site.

One routine postoperative outpatient visit (3 or 6 months): Grip, TUG, HADS, and fee-free InBody (if available).

Postoperative clinical outcomes (e.g., complications within 30 days, length of stay, readmission) are abstracted from the electronic health record per SOP.

Home 6MWT Operating Procedure (app-assisted, summary) Participants are guided to use a flat corridor/sidewalk with markers (e.g., 20-30 m). The app provides standardized instructions (based on ATS principles), a safety checklist (stop for chest pain, severe dyspnea, presyncope), and validity checks (continuous 6 minutes, pause limits, outlier flags). If equipped, step counter or GPS assists distance estimation; otherwise, distance is calculated from marked laps. Adherence (attempts/week, completion %) is automatically captured.

Randomization and Allocation Concealment A centralized, site-stratified, permuted-block sequence is generated by the coordinating center. Allocation is revealed after baseline registration and app onboarding. Because the behavioral nature precludes participant blinding, efforts are made to blind in-hospital outcome assessors (separate staff, standardized scripts, identical test setup).

Data Capture and Management App data are stored under a study ID (no direct identifiers in the app database). On-site measures are entered into an eCRF (secure spreadsheet/EDC with audit trail). Data are backed up on institutional servers with access restricted to authorized study staff. Deidentified analysis datasets are created after data lock. Data retention follows institutional policy and IRB requirements.

Safety and Monitoring Risk is minimal (submaximal walking test and questionnaires). The app includes safety messaging and an emergency stop prompt. Adverse events (AEs) related to testing are recorded; serious AEs are reported per site IRB timelines. A formal independent DMC is not planned due to minimal risk; oversight is provided by the PI and site PIs with periodic monitoring meetings, protocol adherence checks, and query resolution.

Quality Assurance All sites undergo initiation with training on: standardized 6MWT course setup, dynamometer calibration and grip testing posture, TUG instructions/timing, and uniform HADS administration. Checklists are used for each assessment session. The coordinating center performs routine data quality reviews and cross-site consistency checks.

Statistical Considerations (brief) Analyses will follow the intention-to-treat principle. For the prespecified primary endpoint (defined in the Outcome Measures module), between-group comparison will use linear models with adjustment for key covariates (e.g., age, sex, site, surgical category, baseline activity). Secondary outcomes include app-logged adherence, HADS, grip, TUG, fee-free body composition (where available), and postoperative clinical endpoints; these will be analyzed using appropriate generalized linear models. Sensitivity analyses will explore per-protocol effects (e.g., predefined app adherence thresholds). Missing data will be addressed using multiple imputation or model-based methods as appropriate. With 60 participants, the study is powered primarily for feasibility and to estimate effect sizes with reasonable precision to inform future scaling.

Confidentiality and Privacy Only coded study IDs appear in analytical datasets. Contact details are stored separately at the site level. App content avoids collecting unnecessary identifiers. Data transmission uses encrypted channels; access is role-based and logged.

Dissemination Results will be submitted to peer-reviewed journals and scientific meetings. Summary results will be posted on the registry per applicable policies. If effective and feasible, the program is intended to inform broader implementation within ERAS pathways and future larger trials.

Limitations and Mitigation As an open-label behavioral intervention with app logging, performance bias is possible; assessor masking and standardized protocols aim to reduce measurement bias. Fee-free availability of bioimpedance may vary by site; these measures are secondary/exploratory and analyzed accordingly. The design prioritizes feasibility and scalability while preserving rigorous, prespecified endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Elective cancer surgery planned under general anesthesia at a participating site (e.g., gastrointestinal, hepatobiliary-pancreatic, thoracic, gynecologic, or other site-approved cancer operations).
* Ambulatory: able to walk independently (assistive device such as a cane is allowed) and deemed safe to perform a six-minute walk test (6MWT) per investigator judgment.
* Smartphone access and app use: owns/has regular access to a smartphone capable of running the study app and agrees to use the app (notifications, weekly home 6MWT logging, brief daily check-ins).
* Preoperative lead-in: expected interval of ≈14 days or more between consent/randomization and surgery to allow prehabilitation exposure (shorter intervals may be screened but must allow minimum onboarding and at least one home 6MWT).
* Able to understand study procedures and provide written informed consent (Korean or English literacy sufficient to follow app instructions).

Exclusion Criteria:

* Emergency surgery or surgery date that cannot accommodate even minimal prehabilitation onboarding.
* ASA IV or higher, or any unstable/critical condition that, in the investigator's opinion, makes participation unsafe.
* Contraindications to 6MWT/light walking, including but not limited to: unstable angina, recent myocardial infarction (≤30 days), decompensated heart failure, uncontrolled clinically significant arrhythmia, severe symptomatic aortic stenosis, severe uncontrolled pulmonary disease, or investigator-judged safety concerns (e.g., resting severe hypoxemia, high fall risk).
* Non-ambulatory status or musculoskeletal/neurologic conditions that preclude performing a 6MWT.
* Cognitive impairment or psychiatric/behavioral conditions that preclude informed consent or reliable app use.
* Inability or unwillingness to install/use the study app (or lack of regular smartphone access).
* Concurrent enrollment in another interventional clinical trial that would confound outcomes or burden participants (per investigator judgment).
* Any other medical or logistical condition that, in the opinion of the investigator, would interfere with protocol adherence, outcome assessment on the preoperative day, or the routine postoperative follow-up visit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Distance (6MWD) | Preoperative day (within 24-48 hours before surgery)
  Distance in meters covered during a standardized six-minute walk test (6MWT) performed in hospital on the preoperative day. Testing follows ATS-aligned instructions on a marked indoor course (~30 m). Trained staff administer the test and are blinded to group allocation when feasible. The primary endpoint is the absolute distance (meters) on the preoperative day; baseline/home 6MWT collected via the app may be used as a covariate but is not part of the primary measure. Safety prompts (stop for chest pain, severe dyspnea, presyncope) are embedded in the SOP.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS), change | Preoperative day (within 24-48 hours before surgery)
  Change in total HADS score (0-42) from the preoperative day (in-hospital assessment) to the routine postoperative outpatient visit.
Grip strength, change | Preoperative day (within 24-48 hours before surgery)
  Change in maximal hand-grip strength measured with a calibrated dynamometer by trained research staff. Dominant hand is preferred; highest of three trials recorded at each time point.
Timed Up & Go (TUG), change | Preoperative day (within 24-48 hours before surgery)
  Change in time to stand from a chair, walk 3 m, turn, return, and sit. Standardized instructions; best of two trials recorded.
Skeletal muscle mass index (SMI), change | Preoperative day (within 24-48 hours before surgery)
  Change in SMI by bioimpedance analysis (InBody) obtained only via fee-free pathways available at each site; exploratory where not available.
App-logged home 6MWT adherence (preoperative period) | From enrollment to preoperative day (1 day before surgery)
  Percentage of weeks with ≥1 valid home 6-minute walk test (6MWT) logged in the app, per participant, averaged across participants. Validity checks per SOP (continuous 6 minutes, pause limits, outlier flags).
Postoperative complications within 30 days | postoperative day 30
  Number of participants with ≥1 complication graded Clavien-Dindo II or higher, abstracted from the electronic health record per SOP.
hospital length of stay | through study completion, an average of 1 year
  Duration of the index surgical admission.
30-day readmission | postoperative day 30
  Number of participants with all-cause readmission within 30 days of the index discharge.

OTHER OUTCOMES:
App daily check-in completion (preoperative period) | From enrollment to preoperative day (1 day before surgery)
  Percentage of preoperative days with any completed daily check-in (exercise). Averaged across participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided